CLINICAL TRIAL: NCT03211182
Title: Evaluation on Prevention for Metabolic Syndrome and Diabetes Mellitus Through Lifestyle Modification Intervention in Prediabetic Subjects
Brief Title: Lifestyle Modification Intervention in Pre-diabetic Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201110024
Record Dates: First submitted 2017-06-29; First posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: PreDiabetes
Keywords: lifestyle intervention; prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lifestyle intervention group (Experimental): The intervention group was given healthy lifestyle education and individualized counseling by well-trained case manager at baseline, and follow-up phone counseling thereafter.
  Interventions: Behavioral: lifestyle modification intervention
- control group (No Intervention): The control group was given general verbal and written health behavior information to prevent diabetes at baseline without specific individualized advice.

INTERVENTIONS:
Behavioral: lifestyle modification intervention — healthy lifestyle education and individualized counseling by well-trained case manager. The main goals of the lifestyle intervention included regular moderate intensity physical activity 150 min per week or more, and dietary strategies which reduce the risk of developing diabetes. The dietary suggestion was modified by Dietary Approaches to Stop Hypertension (DASH) Diet. Participants with BMI>= 24 kg/m2 were encouraged to gradually lose weight at a rate of 0.5-1.0 kg per week until they achieved a BMI of 24 kg/m2.
  Arms: lifestyle intervention group

SUMMARY:
The lifestyle intervention program focusing on healthy dietary habit and exercise effectively prevents progression to diabetes. Thus, the purpose of this study was to assess the effectiveness of lifestyle intervention program on pre-diabetics subjects in Taiwan.

DETAILED DESCRIPTION:
The study is a 2-parallel groups' randomized controlled trial. Participants with elevated fasting plasma glucose concentrations (FPG 100-125 mg/dl) or glycated hemoglobin (HbA1C 5.7-6.3%) are enrolled. All study subjects are randomized to receive a lifestyle intervention (intervention group) or regular prevention education (control group). The parameters are obtained from physical examination and biochemical assessments by well-trained case manager at baseline and each follow visit (3th months, 6th months and 12th months). All participants complete a structured questionnaire, including basic information, disease history, physical activity, food-frequency, stage of change, and social support situation.

ELIGIBILITY:
Inclusion Criteria:

* 40 years old or over
* elevated fasting plasma glucose concentrations (FPG: 100-125 mg/dl) or glycated hemoglobin(HbA1C: 5.7-6.3%)

Exclusion Criteria:

* having received a diagnosis of diabetes or receiving treatment for diabetes in 3 years
* having a history of cardiovascular disease, stroke, liver disease, kidney disease, cardiopulmonary disease, malignancy or cancer and musculoskeletal impairment
* receiving corticosteroids, androgens, estrogen containing compounds
* who had dietary problem
* pregnant women
* who joined other health intervention study in one year.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-03-07 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
blood sugar | 3 month, 6 month and 12-month follow up
  changes in fasting glucose and glycated hemoglobin

SECONDARY OUTCOMES:
body weight | 3 month, 6 month and 12-month follow up
  weight in kilograms
BMI | 3 month, 6 month and 12-month follow up
  weight and height will be combined to report BMI in kg/m^2
Metabolic syndrome | 3 month, 6 month and 12-month follow up
  defined as 3 or more of 5 components (ie, abdominal obesity, elevated blood pressure, elevated triglycerides, low high-density lipoprotein cholesterol, and dysglycemia)

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yi Chiou, PhD, Study Chair — School of Public Health, Taipei Medical University
Locations (4):
- Taiwan (4):
  - YUANH, Kaohsiung City, Lingya Dist
  - SKH, Taipei, Shilin Dist.
  - TMUH, Taipei, Sinyi District,
  - MMH, Taipei, Zhongshan Dist.

IPD SHARING:
Plan to Share IPD: No